CLINICAL TRIAL: NCT01004367
Title: ACTIVITAL: Health Promotion Intervention in Ecuadorian Adolescents to Promote Healthy Dietary and Physical Activity Patterns.
Brief Title: Health Promotion in Adolescents in Ecuador
Acronym: ACTIVITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); Nutrition Third World, Belgium (Other); VLIR-IUC, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2008/462
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Overweight
Keywords: Promoting healthy lifestyles in adolescents in Ecuador to prevent overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Environmental- and individual based components carried out in the school.
  Interventions: Other: Experimental
- 2 (No Intervention): No intervention

INTERVENTIONS:
Other: Experimental — Environmental- and individual based components carried out in the school.
  Arms: 1

SUMMARY:
Worldwide, low-income and middle-income countries are undergoing rapid demographic and nutritional changes. Populations tend to move from their traditional food habits towards dietary patterns characterized by a more energy-dense diet, while urbanization and technology (work, transport) play a role in the reduction of their physical activity. This shift towards energy-dense diets and lower levels of physical activity are key determinants of chronic diseases. Nowadays, childhood overweight and obesity are becoming a major threat to public health all in low-income and middle-income countries. Clearly, not properly addressing this health problem will only aggravate the already enormous impact of chronic diseases on the social and economic development of these countries. This study aims to develop a culturally relevant school-based prevention intervention among Ecuadorian adolescents (11-13 years old) in Cuenca. The intervention will target behavioural nutrition and physical activity. Intervention strategies will be developed based on theoretical behavioural change models integrated in two complementary frameworks, i.e. (i) the Intervention Mapping protocol, and (ii) the Comprehensive Participatory Planning and Evaluation protocol.

The study includes two phases:

1. A formative research, which will be conducted in order to understand the causality of the school environment and unhealthy eating and low physical activity levels in school-going adolescents, aged 12-13 years old.
2. A paired, cluster-randomized controlled trial including 1400 adolescents (12-13 years old) from 10 pairs of schools (i.e. clusters). Within each pair of clusters, one cluster will be randomly assigned to the intervention and the other to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 11-13 years old
* school-going
* willing to participate

Exclusion Criteria:

* pregnant
* severe medical/physical disorder

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2009-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Behavioural determinants of physical activity and nutrition by determinant questionnaire | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention
Physical activity, physical fitness and sedentarity (questionnaire and accelerometer) | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention
Food intake by 24h recall | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention

SECONDARY OUTCOMES:
Anthropometry | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention
Blood pressure | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention
Socio-economical questionnaire | at 15 and 24 months, additionally, these will be measured 18 months after completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kolsteren, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- Cuenca University, Cuenca, Ecuador

REFERENCES:
- [Derived] Ochoa-Aviles A, Verstraeten R, Huybregts L, Andrade S, Van Camp J, Donoso S, Ramirez PL, Lachat C, Maes L, Kolsteren P. A school-based intervention improved dietary intake outcomes and reduced waist circumference in adolescents: a cluster randomized controlled trial. Nutr J. 2017 Dec 11;16(1):79. doi: 10.1186/s12937-017-0299-5. PMID 29228946
- [Derived] Andrade S, Lachat C, Cardon G, Ochoa-Aviles A, Verstraeten R, Van Camp J, Ortiz J, Ramirez P, Donoso S, Kolsteren P. Two years of school-based intervention program could improve the physical fitness among Ecuadorian adolescents at health risk: subgroups analysis from a cluster-randomized trial. BMC Pediatr. 2016 Apr 22;16:51. doi: 10.1186/s12887-016-0588-8. PMID 27102653
- [Derived] Andrade S, Verloigne M, Cardon G, Kolsteren P, Ochoa-Aviles A, Verstraeten R, Donoso S, Lachat C. School-based intervention on healthy behaviour among Ecuadorian adolescents: effect of a cluster-randomized controlled trial on screen-time. BMC Public Health. 2015 Sep 22;15:942. doi: 10.1186/s12889-015-2274-4. PMID 26395439
- [Derived] Andrade S, Lachat C, Ochoa-Aviles A, Verstraeten R, Huybregts L, Roberfroid D, Andrade D, Camp JV, Rojas R, Donoso S, Cardon G, Kolsteren P. A school-based intervention improves physical fitness in Ecuadorian adolescents: a cluster-randomized controlled trial. Int J Behav Nutr Phys Act. 2014 Dec 10;11:153. doi: 10.1186/s12966-014-0153-5. PMID 25490946